CLINICAL TRIAL: NCT05176119
Title: The Effect of Low Dose Nalbuphine or Ketamine in the Prevention of Emergence Agitation After Sevoflurane Anesthesia in Children Undergoing Tonsillectomy With or Without Adenoidectomy
Brief Title: Nalbuphine Versus Ketamine for Prevention of Emergence Agitation After Sevoflurane in Children Undergoing Tonsillectomy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Diaaeldein Mahmoud Haiba, Lecture of Anesthesia, ICU & Pain mangement faculty od medicine, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: MS 160/2021
Record Dates: First submitted 2021-10-19; First posted 2022-01-04 (Actual); Last update posted 2022-01-04 (Actual); Status verified 2021-12

CONDITIONS: Pediatric ALL; Pediatric Anesthesia
Keywords: Emergence agitation; Ketamine; Nalbuphine; Sevoflurane.
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Emergence Delirium | interventions — Nalbuphine; Ketamine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Nalbuphine arm (Active Comparator): 0.1 mg /kg nalbuphine was given to 30 patients
  Interventions: Drug: Nalbuphine Injection
- Ketamine arm (Active Comparator): 0.25 mg /kg ketamine was given to 30 patients
  Interventions: Drug: Ketamine
- Saline arm (Placebo Comparator): an equivalent volume of normal saline was given to 30 patients
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Nalbuphine Injection — At the end of the surgery and just before discontinuation of sevoflurane and extubation the study medications will be prepared by the local pharmacy as 10 ml syringes that were handed to the anesthesiologist in charge in OR room who was blinded to the nature of the medications.
  Arms: Nalbuphine arm
Drug: Ketamine — At the end of the surgery and just before discontinuation of sevoflurane and extubation the study medications will be prepared by the local pharmacy as 10 ml syringes that were handed to the anesthesiologist in charge in OR room who was blinded to the nature of the medications.
  Arms: Ketamine arm
Drug: Saline — At the end of the surgery and just before discontinuation of sevoflurane and extubation the study medications will be prepared by the local pharmacy as 10 ml syringes that were handed to the anesthesiologist in charge in OR room who was blinded to the nature of the medications.
  Arms: Saline arm

SUMMARY:
The effect of low dose nalbuphine or ketamine in the prevention of emergence agitation after sevoflurane anesthesia in children undergoing tonsillectomy with or without adenoidectomy.

This randomized double-blind study was carried out at, Ain shams University Hospitals, from March 2021 to June 2021 on 90 patients after approval of the ethical committee.

DETAILED DESCRIPTION:
Emergence agitation (EA) in children is increased after sevoflurane anesthesia. Nalbuphine and midazolam have been used for prophylactic treatment with controversial results.

Patients and Methods:Totally, 90 children between 4 and 10 years of age and of American Society of Anesthesiologists I-II undergoing adenotonsillectomy under sevoflurane-based anesthesia were enrolled in the study. Children were randomly allocated to one of the three groups: Group N received nalbuphine 0.1 mg/kg, Group K received ketamine 0.25 mg /kg and Group S received the equivalent volume saline. The study medications was given after discontinuation of sevoflurane by the end of surgery. In the post anesthesia care unit emergence agitation was assessed with emergence agitation scale upon admission (T0), after 5 min (T5), 10 min (T10), 15 min (T15), 20 min (T20), 25 min (T25) and 30 min (T30).

ELIGIBILITY:
Inclusion Criteria:

Pediatric patients undergoing tonsillectomy with or without adenoidectomy

1. Age 4 - 10 years.
2. Sex: Both sexes
3. Patients with ASA classificaion I and II.

Exclusion Criteria:

1. Declining to give written informed consent.
2. History of allergy to the medications used in the study.
3. psychiatric disorder.
4. ASA classification III-V.
5. Fever ,cough , asthma or upper respiratory tract infection .
6. Anticipated difficult airway .
7. Hearing defect .
8. Neurological disorder.
9. Family history of malignant hyperthermia .

Ages: 4 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Actual)
Dates: Start 2021-03-25 (Actual); Primary Completion 2021-06-25 (Actual); Study Completion 2021-06-25 (Actual)

PRIMARY OUTCOMES:
Emergence Agitation | At Time zero (The time of extubation)
  5 step Emergence Agitation scale: describing change in mental status of the children during emergence from general anesthesia. The minimum value is 1 and maximum value is 5, and higher scores mean a better outcome.
  Score 1 Obtunded with no response to stimulation. Score 2 Asleep but responsive to movement or stimulation Score 3 Awake and responsive Score 4 Crying Score 5 Thrashing behaviour that requires restraint

SECONDARY OUTCOMES:
Emergence Agitation at post anesthesia care unit(PACU) | At time of delivery to PACU
  5 step Emergence Agitation scale: describing change in mental status of the children during emergence from general anesthesia. The minimum value is 1 and maximum value is 5, and higher scores mean a better outcome.
  Score 1 Obtunded with no response to stimulation. Score 2 Asleep but responsive to movement or stimulation Score 3 Awake and responsive Score 4 Crying Score 5 Thrashing behaviour that requires restraint
Post-operative pain | 30 minutes
  Occurrence of post-operative pain using Modified Children's Hospital of Eastern Ontario Pain Scale (mCHEOPS). It is a behavioral observational Pain Scale for evaluating postoperative pain in young children. It can be used to monitor the effectiveness of interventions for reducing the pain and discomfort. The minimum value is 0 and maximum value is 10, and higher scores mean a worse condition.
Midazolam given for emergence agitation | 30 minutes
  It is described as given or not given.
Duration in PACU | 45 minutes
  duration from receiving the patient in the post anaesthesia care unit till discharge to the ward.it described in the form of minutes.
Time to hospital discharge. | 6 hours
  Duration from receiving the patient in the post anesthesia care unit till hospital discharge.it described in the form of hours.
Occurrence of postoperative nausea and vomiting | 120 minutes
  described in the from of occurred or not occurred
Occurrence of laryngeal spasm | 120 minutes
  described in the from of occurred or not occurred
Post-tonsillectomy bleeding. | 120 minutes
  described in the from of occurred or not occurred

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams university hospitals, Cairo, Al Abbassia, Egypt

IPD SHARING:
Plan to Share IPD: No